CLINICAL TRIAL: NCT06594432
Title: A Study on the Efficacy and Safety of Molecular Subtype-Guided R-CHOP-MTX±Zanubrutinib Treatment in Newly Diagnosed DLBCL Patients with Central Nervous System Involvement
Brief Title: Molecular Subtype-Guided R-CHOP-MTX±Zanubrutinib Treatment in Newly Diagnosed DLBCL Patients with Central Nervous System Involvement
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, Principal Investigator, The First Affiliated Hospital with Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-433
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MCD, BN2, and N1 subtypes (Other)
  Interventions: Drug: R-CHOP+Z+MTX
- EZB, A53, and other gene subtypes (Other)
  Interventions: Drug: R-CHOP+MTX

INTERVENTIONS:
Drug: R-CHOP+Z+MTX — After receiving 1 cycle of pre-treatment with the R-CHOP regimen, patients with CSF-ctDNA (+) and MCD, BN2, and N1 subtypes will receive 5 cycles of R-CHOP combined with MTX + Zanubrutinib, followed by 1 cycle of R-MTX-Zanubrutinib.
  After completing the above induction therapy, Patients with negative CSF-ctDNA results will continue with one more cycle of Rituximab. For patients with positive CSF-ctDNA results, the investigator will decide to continue treatment with Rituximab one more cycle combined with Temozolomide, Pomalidomide, or Lenalidomide, etc., until CSF-ctDNA turns negative.
  Each combined regimen consists of a 21-day treatment cycle, and efficacy will be evaluated every three treatment cycles.
  Arms: MCD, BN2, and N1 subtypes
Drug: R-CHOP+MTX — After receiving 1 cycle of pre-treatment with the R-CHOP regimen, patients with CSF-ctDNA (+) and EZB, A53, and other gene subtypes will receive 5 cycles of R-CHOP combined with MTX, followed by 1 cycle of R-MTX.
  After completing the above induction therapy, Patients with negative CSF-ctDNA results will continue with one more cycle of Rituximab. For patients with positive CSF-ctDNA results, the investigator will decide to continue treatment with Rituximab one more cycle combined with Temozolomide, Pomalidomide, or Lenalidomide, etc., until CSF-ctDNA turns negative.
  Each combined regimen consists of a 21-day treatment cycle, and efficacy will be evaluated every three treatment cycles.
  Arms: EZB, A53, and other gene subtypes

SUMMARY:
Evaluate the Efficacy and Safety of R-CHOP-MTX±Zanubrutinib in Newly Diagnosed Diffuse Large B-Cell Lymphoma Patients with Central Nervous System Involvement, and Explore the Efficacy Indicators of CSF-ctDNA.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤80 years, regardless of gender;
2. Patients with pathologically confirmed, previously untreated diffuse large B-cell lymphoma (DLBCL) who are CSF-ctDNA positive for secondary CNS lymphoma (SCNSL);
3. MRI or CT of the brain showing substantial lesions in the central nervous system; patients with only meningeal lesions must have CSF cytology confirming lymphoma cells and/or imaging findings consistent with CSF examination;
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-3;
5. Organ function levels meeting the following requirements:Absolute neutrophil count ≥1.5×10^9/L, platelets ≥75×10^9/L, hemoglobin ≥90g/L (if bone marrow is involved, platelets ≥50×10^9/L).
6. Liver function: ALT and AST ≤2.5 times the upper limit of normal, total bilirubin ≤2 times the upper limit of normal.

8.Renal function: creatinine ≤1.5 times the upper limit of normal; creatinine clearance rate ≥40 ml/min (assessed according to the Cockcroft-Gault formula or the estimated glomerular filtration rate [eGFR] from the Modification of Diet in Renal Disease [MDRD] formula).

9.Coagulation function: International Normalized Ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5×ULN.

10.Expected survival time >3 months; 11.No radiotherapy, chemotherapy, or antibody therapy within 3 weeks before medication; no targeted therapy within 10 days before medication; 12.Female subjects of childbearing potential must agree to use effective contraception during the study and for at least 90 days after the last dose of the study drug. Male subjects must be sterilized, i.e., vasectomy, or use barrier methods, while their female partners use the aforementioned effective contraception.

13.Signed written informed consent before trial screening.

Exclusion Criteria:

1. Previous treatment with BTK inhibitors;
2. Received targeted therapy within 10 days before starting the study drug, or systemic chemotherapy, radiotherapy, or antibody therapy within 3 weeks before starting the study drug;
3. Abnormal liver function (total bilirubin >2 times the normal value, ALT or AST >2.5 times the normal value), abnormal renal function (serum creatinine >1.5 times the normal value);
4. Currently have clinically significant active cardiovascular disease, such as uncontrolled arrhythmias, congestive heart failure, any grade 3 or 4 heart disease as determined by the New York Heart Association (NYHA) functional classification, or a history of myocardial infarction within 6 months before screening;
5. QTcF >450 msecs or other significant ECG abnormalities, including second-degree type II atrioventricular (AV) block or third-degree AV block;
6. Previous chemotherapy with unresolved toxicity (toxicity not resolved to ≤ grade 1 according to NCI-CTCAE 5.0, except for alopecia, absolute neutrophil count (ANC), and platelets);
7. Patients with active bleeding;
8. Patients with active infections or persistent fever within 14 days before enrollment (excluding tumor-related fever);
9. Patients with active HBV, HCV, and HIV infections;
10. Patients with serous cavity effusion;
11. Patients who have not completed 4 weeks after major organ surgery;
12. Patients receiving strong inhibitors or strong inducers of cytochrome P450 family 3 subfamily A (CYP3A);
13. Pregnant or lactating women and patients of childbearing potential who are unwilling to use contraception;
14. Patients with mental disorders/unable to obtain informed consent;
15. Patients who abuse drugs or have long-term alcoholism that affects the evaluation of trial results;
16. Patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
CSF-ctDNA negativity rate at the end of induction therapy (EOT) | At the end of induction therapy (EOT), an average of 6 months

SECONDARY OUTCOMES:
Progression Free Survival（PFS） | 2 years
Complete Response Rate（CR） | End of treatment visit (after last dose of Cycle 7 [Cycle length=21 days]）
Overall Survival（OS） | up to approximately 24 months
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From enrollment to study completion, a maximum of 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, Principal Investigator — The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital)
Locations (1):
- Hematological Department, People's Hospital of Jiangsu Province, Nanjing, Jiangsu, China